CLINICAL TRIAL: NCT01770535
Title: A Single-Centre Prospective Phase 0 Translational Study for Predicting Response of High Grade Serous Ovarian Cancers to Paclitaxel Chemotherapy
Brief Title: Oxford Ovarian Cancer Predict Chemotherapy Response 01
Acronym: OXO-PCR-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OXO-PCR-01
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer, paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ovarian cancer biopsy tissue samples Eyebrow hair follicles Blood samples Surgical tissue samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to understand why there are differences between individuals in the way they respond to paclitaxel chemotherapy.

DETAILED DESCRIPTION:
While paclitaxel is very effective in killing cancer cells in a proportion of patients, some patients don't respond to this treatment. As with any chemotherapy, paclitaxel is associated with unpleasant side effects. We are doing this study to try and understand what is happening in cancer cells in different individuals after paclitaxel treatment that make them respond differently to the same treatment. We hope that this study will enable us to develop a method to identify women who are suitable for this form of treatment. We also want to understand why some cancer cells don't get killed with paclitaxel. This information will help us to select treatment to suit an individual patient, and thus improve the outcome of treatment and avoid giving treatment that will not benefit the patient.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years of age
* Newly diagnosed and histology confirmed primary high grade serous ovarian cancer, high grade serous fallopian tube cancer and primary peritoneal carcinoma.
* Radiological and laparoscopic confirmation of FIGO stage 3C or 4 ovarian cancer.
* Radiological evidence of omental or peritoneal deposits that are accessible for radiology-guided biopsy.
* At least one lesion on CT scan measuring at least 2 cm in maximum diameter performed in the past 31 days. Slightly older scans may be accepted at the discretion of the CI providing the results are considered to remain clinically relevant.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Life expectancy of at least 6 months.
* The patient is willing and able to provide written informed consent and comply with the protocol for the duration of the study, and scheduled visits and examinations.
* Acceptable haematological and biochemical indices

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological and histological evidence of advanced ovarian cancer, who would standardly be managed by primary chemotherapy and interval debulking surgery
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between βIII tubulin expression and Mitotic Index (MI) following single agent paclitaxel treatment | Before and 24-hours after paclitaxel treatment
  Correlation between βIII tubulin expression and Mitotic Index (MI) before and after single agent paclitaxel treatment to determine whether overexpression of βIII tubulin is associated with Paclitaxel resistance

SECONDARY OUTCOMES:
Correlation between mitotic index and the magnitude of CA125 response | three weeks after paclitaxel treatment
  Correlation between mitotic index and the magnitude of CA125 response will be analysed to investigate whether post-paclitaxel mitotic index is a determinant of clinical response in ovarian cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Churchill Hospital, Oxford, United Kingdom